CLINICAL TRIAL: NCT01436149
Title: The SPD489-322 Phase 3, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Flexible Dose Titration, Efficacy and Safety Study of SPD489 in Combination With an Antidepressant in the Treatment of Adults With Major Depressive Disorder With Inadequate Response to Prospective Treatment With an Antidepressant
Brief Title: Efficacy and Safety Study of SPD489 in Combination With an Antidepressant in the Treatment of Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-322; 2011-003018-17 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Antidepressant + SPD489 (Experimental)
  Interventions: Drug: SPD489 (Lisdexamfetamine dimesylate )
- Antidepressant + Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 (Lisdexamfetamine dimesylate ) — Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride) oral, once daily + SPD489 (oral, 20, 30, 50 or 70 mg, once daily) for 8 weeks
  Other Names: Vyvanse
  Arms: Antidepressant + SPD489
Drug: Placebo — Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride) oral, once daily + Placebo (oral, once daily) for 8 weeks
  Arms: Antidepressant + Placebo

SUMMARY:
This study will examine SPD489 in subjects aged 18-65 with major depressive disorder (MDD) who are taking certain types of antidepressants but continue to have residual depression symptoms. Eligible patients will remain on their antidepressant but will be randomized to either receive supplemental SPD489 or placebo (i.e. sugar pill). The purpose of this study is to help answer the following questions:

* How safe is SPD489 for the supplemental treatment of depression and what are the side effects that might be related to it?
* Can supplemental SPD489 help patients who still have residual depression symptoms while taking an antidepressant?
* How much SPD489 should be given to patients with depression who are also taking an antidepressant?
* How does SPD489 compare to placebo in depressed patients who are also taking an antidepressant?

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide written, personally signed, and dated informed consent to participate in the study.
* Subject is between 18 and 65 years of age.
* Subject has a primary diagnosis of non-psychotic MDD (single or recurrent).
* Subject has a MADRS total score 24.
* Subject who is female, must have a negative serum beta human chorionic gonadotropin (HCG) pregnancy test and a negative urine pregnancy test at the and agrees to comply with any applicable contraceptive requirements of the protocol.
* Subject is able to swallow a capsule.

Exclusion Criteria:

* Subject whose current episode of MDD has not responded to an adequate treatment regimen with 2 or more approved single antidepressant agents.
* Subject who has a lifetime history of treatment resistant depression.
* Subject has a current co-morbid psychiatric disorder. Excluded are: any significant Axis II disorder (including borderline personality disorder), any bipolar disorder, any current or lifetime psychosis, post traumatic stress disorder, obsessive compulsive disorder, any pervasive development disorder, anorexia nervosa and bulimia nervosa.
* Subject has been hospitalized (within the last 12 months) for their current MDD episode.
* Subject has a current or lifetime history of attention-deficit/hyperactivity disorder (ADHD).
* Subject has a first degree relative that has been diagnosed with bipolar I disorder.
* Subject has a recent history (within the last 6 months) of suspected substance abuse or dependence disorder
* Subject is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt within the past 3 years, or is currently demonstrating active suicidal ideation.
* Subject has a concurrent chronic or acute illness or unstable medical condition.
* Subject has a history of seizures (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder, serious neurological disease, history of significant head trauma, dementia, cerebrovascular disease, Parkinson's disease, or intracranial lesions.
* Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems.
* Subject has a history of thyroid disorder that has not been stabilized on thyroid medication or treatment within 3 months prior to the Screening Visit.
* Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
* Subject has glaucoma.
* Subject has a history of moderate to severe hypertension.
* Current use of any other medications (including over-the-counter [OTC], herbal or homeopathic preparations) that have central nervous system effects.
* Subject has had electroconvulsive therapy (ECT) for the current depressive episode 3 months prior.
* The subject has a known or suspected intolerance, hypersensitivity, or contraindications to their assigned antidepressant treatments (escitalopram oxalate, sertraline HCl, venlafaxine HCl extended release, or duloxetine HCl).
* Subject has a positive urine drug result.
* Subject has a body mass index (BMI) of <18.5 or >40.
* Subject is female and is pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1262 (Actual)
Dates: Start 2011-10-27 (Actual); Primary Completion 2013-12-23 (Actual); Study Completion 2013-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (85):
- United States (47):
  - Birmingham Research Group, Birmingham, Alabama
  - AV Institue, Inc., Carson, California
  - University of California, Irvine Child Development Center, Irvine, California
  - South Coast Clinicals, Norwalk, California
  - North County Clinical Research, Oceanside, California
  - Pasadena Research Institute, LLC, Pasadena, California
  - Affiliated Research Institute, San Diego, California
  - Clinical Innovations, Inc., San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Geriatric and Adult Psychiatry, LLC, Hamden, Connecticut
  - Middlexex Hospital Center for Behavioral Health, Middletown, Connecticut
  - CNS Clinical Research Group, Coral Springs, Florida
  - Emerald Coast Mood & Memory, PA, Fort Walton Beach, Florida
  - Florida Clinical Research Center, LLC., Maitland, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Compass Research, LLC, Orlando, Florida
  - Meridien Research, St. Petersburg, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Carman Research, Smyrna, Georgia
  - American Medical Research, Inc., Oak Brook, Illinois
  - The Davis Clinic, Indianapolis, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - MCM Clinical Research LLC, Florence, Kentucky
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Potomac Grove Clinical Research Center, Gaithersburg, Maryland
  - Office of Marc Hertzman, MD, Rockville, Maryland
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Bioscience Research, LLC, Mount Kisco, New York
  - Fieve Clinical Research, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Triangle Neuropsychiatry, Durham, North Carolina
  - Rcihard H. Weisler, MD, PA & Associates, Raleigh, North Carolina
  - Community Research, Cincinnati, Ohio
  - Lindner Center of HOPE, Mason, Ohio
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - CRI Worldwide LLC, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Summit Research Network (Seattle) LLC, Seattle, Washington
- Canada (20):
  - Dr. Alexander McIntyre Inc, Penticton, British Columbia
  - Dr. D. McIntosh & Dr. K. Kjernisted Clinical Research Inc., Vancouver, British Columbia
  - Aggarwal & Associates Ltd., Brampton, Ontario
  - Depression, Mood Disorders and Schizophrenia Treatment Centre, Burlington, Ontario
  - Chatham-Kent Clinical Trials Research Center, Chatham, Ontario
  - Regional Mental Health Care, London, Ontario
  - Anxiety and Mood Disorder Center, Mississauga, Ontario
  - Medical Research Associates, Mississauga, Ontario
  - A.K. Karan Holdings, Oakville, Ontario
  - International Sleep Clinic, West Parry Sound Health Centre, Parry Sound, Ontario
  - START Clinic for Mood and Anxiety Disorders, Toronto, Ontario
  - Univ Health Network, Toronto Western Hospital, Toronto, Ontario
  - Sleep & Alertness Clinic (Sleep & Alertness Research, Inc.), Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Windsor Regional Hospital-Tayfour Campus, Windsor, Ontario
  - Pierre-Janet Hospital, Gatineau, Quebec
  - l'Hopital Louis H. Lafontaine, Montreal, Quebec
  - Kells Medical Research Group Inc., Pointe-Claire, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - Q&T Research Sherbrooke, Sherbrooke, Quebec
- Croatia (2):
  - Poliklinika Neuron, Zagreb
  - Psychiatric Clinic Vrapoe, Zagreb
- Mexico (5):
  - Centro Regiomontano de Investigacion S.C. (CRI), Monterrey, Nuevo León
  - Hospital Aranda de la Parra, León
  - Instituto de Infromacion e Investigación en Salud Mental (INFOSAME), Nuevo León
  - Consultorio Especializado en Psiquiatria Infantil y Adolescentes, San Luis Potosí City
  - B & B Investigaciones Medicas S.C., Sinaloa
- Puerto Rico (2):
  - Dharma Institute & Research Center, San Juan
  - INSPIRA Clinical Research, San Juan
- Spain (9):
  - Hospital de la Santa Creo l Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Servicio de Psiquiatria, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Fundacion de Alcorcon, Madrid
  - Hospital Universitario de Henares, Madrid
  - Centro de Salud Mental Il la Corredoria, Oviedo
  - Centro Salud Alamedilla Unidad de Salud Mental, Salamanca
  - Complejo hospitalario de Zamora, Zamora
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Result] Richards C, McIntyre RS, Weisler R, Sambunaris A, Brawman-Mintzer O, Gao J, Geibel B, Dauphin M, Madhoo M. Lisdexamfetamine dimesylate augmentation for adults with major depressive disorder and inadequate response to antidepressant monotherapy: Results from 2 phase 3, multicenter, randomized, double-blind, placebo-controlled studies. J Affect Disord. 2016 Dec;206:151-160. doi: 10.1016/j.jad.2016.07.006. Epub 2016 Jul 5. PMID 27474961

RESULTS

PARTICIPANT FLOW:
Groups:
- Antidepressant + Single-blind Placebo: Subjects received unblinded oral, once daily standard antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended-release, or duloxetine hydrochloride) plus oral, once daily placebo (matching SPD489).
- Antidepressant + Double-blind Placebo: Subjects received assigned oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) plus oral, once daily, double-blind placebo (matching SPD489).
- Antidepressant + Double-blind SPD489: Subjects received assigned oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) plus oral, once daily SPD489 (Lisdexamfetamine dimesylate optimized among 20, 30, 50, or 70 mg dose).
Period: Antidepressant Lead-in Phase
Arm/Group | Antidepressant + Single-blind Placebo | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489
Started | 1262 (Twenty-three subjects were enrolled but not dosed.) | 0 | 0
Completed | 896 | 0 | 0
Not Completed | 366 | 0 | 0
Not completed — Adverse Event | 39 | 0 | 0
Not completed — Protocol Violation | 29 | 0 | 0
Not completed — Withdrawal by Subject | 61 | 0 | 0
Not completed — Lost to Follow-up | 96 | 0 | 0
Not completed — Met BP Or Pulse Withdrawal Criteria | 22 | 0 | 0
Not completed — Other | 119 | 0 | 0
Period: Randomized Phase
Arm/Group | Antidepressant + Single-blind Placebo | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489
Started | 492 (These subjects were not included in the Safety Analysis Set or Full Analysis Set.) | 202 (One subject did not receive at least 1 dose of double-blind treatment.) | 202 (One subject did not receive at least 1 dose of double-blind treatment.)
Completed | 415 | 164 | 160 (1 subject completed the study without a Visit 14 MADRS and was not included in the completers set.)
Not Completed | 77 | 38 | 42
Not completed — Adverse Event | 9 | 10 | 11
Not completed — Protocol Violation | 4 | 5 | 0
Not completed — Withdrawal by Subject | 16 | 10 | 10
Not completed — Lost to Follow-up | 34 | 5 | 6
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Met BP Or Pulse Withdrawal Criteria | 2 | 3 | 3
Not completed — Other | 12 | 5 | 11

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects who took at least 1 dose of randomized investigational product and who had at least 1 safety assessment (e.g., coming back for any visit, reporting of an adverse event [AE], or reporting the absence of AEs) after the Augmentation Baseline Visit (Visit 8).
Groups:
- Antidepressant + Double-blind Placebo: Oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) plus oral, once daily, double-blind placebo (matching SPD489) for 8 weeks.
- Antidepressant + Double-blind SPD489: Oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) plus oral, once daily SPD489 (Lisdexamfetamine dimesylate optimized among 20, 30, 50, or 70 mg dose) for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 | Total
Number analyzed (Participants) | 201 | 201 | 402
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (12.04) | 42.2 (12.32) | 42 (12.17)
Age, Customized [Count of Participants; unit: Participants]
  18-55 years | 173 | 170 | 343
  56-65 years | 28 | 31 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 129 | 262
  Male | 68 | 72 | 140

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at up to 8 Weeks
Description: MADRS is a validated, 10-item rating scale with each item being scored on a scale from 0-6 with a total score ranging from 0-60. Lower scores indicate a decreased severity of depression.
Time Frame: 8 weeks
Population: Full Analysis Set: Subjects who took at least 1 dose of randomized investigational product and who had at least 1 valid primary efficacy measurement of the MADRS total score after the Augmentation Baseline Visit (Visit 8).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Antidepressant + Placebo: Antidepressant + Placebo: Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) oral, once daily + Placebo (oral, once daily) for 8 weeks.
- Antidepressant + SPD489: Antidepressant + SPD489 (Lisdexamfetamine dimesylate): Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) oral, once daily + SPD489 (optimized as a 20, 30, 50, or 70 mg dose, oral, once daily), for 8 weeks.
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 200 | 200
units on a scale | -6.3 [-7.6 to -4.9] | -6.1 [-7.5 to -4.8]
Statistical Analysis 1: Comparison: Antidepressant + Placebo vs Antidepressant + SPD489; Test type: Superiority or Other; p = 0.883, Mixed- effects Model for Repeat Measures; Difference in LS Mean = 0.1, 95% CI 2-sided [-1.7 to 2.0], Standard Error of Mean 0.96

2. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at up to 8 Weeks
Description: Designed to evaluate the extent to which illness symptoms impact a subject's life in 3 areas: work/school, social, and family/home. Each area is scored on a scale from 0 (no impairment) to 10 (highly impaired) with a total score ranging from 0 (unimpaired) to 30 (highly impaired). Lower scores translate into less impairment.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 200 | 200
units on a scale | -4.3 [-5.3 to -3.3] | -4.7 [-5.6 to -3.7]
Statistical Analysis 1: Comparison: Antidepressant + Placebo vs Antidepressant + SPD489; Test type: Superiority or Other; p = 0.576, Mixed- effects Model for Repeat Measures; Difference in LS Mean = -0.4, 95% CI 2-sided [-1.8 to 1.0], Standard Error of Mean 0.69

3. Secondary Outcome: Percentage of Participants Achieving a 25% Response on the MADRS
Description: The percentage of subjects who achieved a 25% response (i.e., ≥25% reduction in MADRS total score from Lead-in Baseline, Visit 2; Week 0). A comparison was performed at Visit 14/Early Termination (ET) (Week 16/ET).
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 200 | 200
percentage of participants | 65.0 | 74.5

4. Secondary Outcome: Percentage of Participants Achieving a 50% Response on the MADRS
Description: The percentage of subjects who achieved a 50% response (i.e., ≥50% reduction in MADRS total score from Lead-in Baseline, Visit 2; Week 0). A comparison was performed at Visit 14/ET (Week 16/ET).
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 200 | 200
percentage of participants | 38.5 | 41.0

5. Secondary Outcome: Percentage of Participants Achieving Remission on the MADRS
Description: MADRS remission was defined as a MADRS total score of ≤10. A comparison was performed at Visit 14/ET (Week 16/ET).
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 200 | 200
percentage of participants | 22.5 | 18.5

6. Secondary Outcome: Mean Change From Baseline Over Time in MADRS Total Score
Description: as for outcome 1
Time Frame: Baseline and up to 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 200 | 200
units on a scale
  Visit 9 (Week 9) | -2.2 [-3.1 to -1.2] | -3.4 [-4.3 to -2.4]
  Visit 10 (Week 10) | -3.8 [-4.9 to -2.7] | -4.2 [-5.3 to -3.2]
  Visit 11 (Week 11) | -6.0 [-7.2 to -4.8] | -5.4 [-6.6 to -4.2]
  Visit 12 (Week 12) | -6.2 [-7.4 to -5.0] | -5.6 [-6.8 to -4.4]
  Visit 13 (Week 14) | -7.4 [-8.7 to -6.0] | -7.3 [-8.6 to -6.0]
  Visit 14 (Week 16) | -6.3 [-7.6 to -4.9] | -6.1 [-7.5 to -4.8]

7. Secondary Outcome: Mean Change From Baseline in the Quick Inventory of Depressive Symptomatology - Self Report (QIDS SR)
Description: The QIDS-SR is a self-administered questionnaire designed to rate depressive symptoms. The scale contains 16 items, each scored using a 4-point scale ranging from 0 (representing the most favorable response [low amount of symptom]) to 3 (representing the least favorable response [frequent/intense symptom]). The total score could range from 0 (no depression) to 27 (very severe depression). Higher scores represent more severe depressive symptoms.
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 186 | 185
units on a scale | -2.6 [-3.2 to -1.9] | -2.3 [-2.9 to -1.7]

8. Secondary Outcome: Mean Change From Baseline in the Short Form-12 Health Survey V2 (SF-12V2)
Description: Total score ranges from 0 (lowest level of health) - 100 (highest level of health) on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability (i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability). Higher scores are associated with better quality of life.
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 189 | 186
units on a scale
  Physical | 0.69 [-0.39 to 1.77] | -0.81 [-1.89 to 0.28]
  Mental | 5.59 [3.93 to 7.25] | 6.5 [4.84 to 8.16]

9. Secondary Outcome: Mean Change From Baseline in the Quality of Life Enjoyment Satisfaction Questionnaire Short Form (Q-LES-Q-SF)
Description: The short form is a 16-item self-report questionnaire which evaluates general subject satisfaction with health, mood, relationships, functioning in daily life, and the treatment being taken. Overall level of satisfaction is evaluated on a 5-point scale from 1 (very poor) to 5 (very good). The total score ranges from 14-70 (last two items on the form are not included in the total score). A higher score indicates a better quality of life.
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 188 | 184
units on a scale | 7.2 [4.9 to 9.5] | 7.0 [4.7 to 9.3]

10. Secondary Outcome: Clinical Global Impressions - Global Improvement (CGI-I)
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 199 | 199
percentage of participants
  Improved | 53.3 | 55.3
  Not Improved | 46.2 | 44.7
  Not Assessed | 0.5 | 0

11. Secondary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred. The assessment is done by the nature of the responses, not by a numbered scale.
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 201 | 201
percentage of participants
  ≥1 postive suicidal ideation | 7.0 | 7.0
  ≥1 suicidal attempt | 0.5 | 0

12. Secondary Outcome: Amphetamine Cessation Symptom Assessment (ACSA)
Description: ACSA scale has 16 symptom items rated on a scale from 0 (not at all) to 4 (extremely) with a possible total score range of 0 to 64. Higher scores indicate greater withdrawal symptom severity.
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Number analyzed (Participants) | 178 | 183
units on a scale | 15.1 (10.71) | 14.7 (10.94)

ADVERSE EVENTS:
Groups:
- Antidepressant + Placebo: Oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) plus oral, once daily, double-blind placebo (matching SPD489).
- Antidepressant + SPD489: Oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride), plus oral, once daily SPD489 (Lisdexamfetamine dimesylate optimized among 20, 30, 50 or 70 mg dose).
Arm/Group | Antidepressant + Placebo | Antidepressant + SPD489
Serious Adverse Events (participants affected / at risk) | 5/201 | 3/201
Other Adverse Events (participants affected / at risk) | 54/201 | 70/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant + Placebo (N=201) | Antidepressant + SPD489 (N=201)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant + Placebo (N=201) | Antidepressant + SPD489 (N=201)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 19 (19)
Nausea (Gastrointestinal disorders) | 10 (11) | 13 (13)
Nasopharyngitis (Infections and infestations) | 4 (4) | 11 (12)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 15 (17)
Headache (Nervous system disorders) | 21 (28) | 13 (14)
Insomnia (Psychiatric disorders) | 15 (16) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.